CLINICAL TRIAL: NCT02751710
Title: Impact of 18F-FDG PET-CT Versus Conventional Staging in the Management of Patients Presenting With Clinical Stage III Breast Cancer
Acronym: PET ABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Cancer Care Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OCOG-2016-PETABC
Record Dates: First submitted 2016-04-15; First posted 2016-04-26 (Estimated); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Stage III Breast Cancer (T0N2, T1N2, T2N2, T3N1, 2 or T4); Stage IIb Breast Cancer (T3N0)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole-body FDG PET-CT alone (Experimental)
  Interventions: Other: Whole-body FDG PET-CT alone
- Conventional breast cancer staging (No Intervention): Conventional breast cancer staging consisting of a bone scan and CT imaging with contrast of the chest / abdomen & pelvis

INTERVENTIONS:
Other: Whole-body FDG PET-CT alone — FDG PET-CT imaging
  Arms: Whole-body FDG PET-CT alone

SUMMARY:
This trial is being conducted to determine the impact of whole body FDG PET-CT vs. conventional staging in the management of patients presenting with clinical Stage III breast cancer. Eligible consenting patients with ductal or mixed histology breast cancer will be randomized 1:1 to whole body FDG PET-CT or conventional staging. Eligible consenting patients with lobular only histology will be entered into a separate single arm prospective study and will undergo whole body FDG PET-CT, CT with contrast of the chest/abdomen & pelvis and a bone scan.

ELIGIBILITY:
Inclusion Criteria:

* Women (or men) with histological evidence of breast cancer for whom potentially curative treatment is planned.
* Based on clinical information (physical exam, imaging):

  1. Stage III breast cancer (T0N2, T1N2, T2N2, T3N1, 2 or T4), or
  2. Stage IIb breast cancer (T3N0), Note: T2N1 is not eligible
* Considered for combined modality therapy (surgical resection, chemotherapy, radiotherapy) of curative intent.

Exclusion Criteria:

* Age < 18 years,
* ECOG performance status > and = 3,
* Prior systemic therapy (e.g. neo-adjuvant chemotherapy or hormonal therapy) for current breast cancer,
* Previous staging investigations for current breast cancer,
* Breast cancer with primary histological subtypes other than ductal or lobular (Note: Patients with mixed disease will be eligible for randomization),
* Clinical suspicion of metastatic disease,
* Relative contraindications to PET (e.g. uncontrolled diabetes (i.e. inability to decrease serum glucose below 10.2 mmol/L), claustrophobia, inability to be still for 30 minutes),
* Inability to lie supine for imaging with PET-CT,
* Inability to undergo CT because of known allergy to contrast,
* History of another invasive malignancy within the previous two years (exception of non melanoma skin cancer) or a synchronous primary cancer, including a synchronous contralateral breast cancer (Note: Patients found to have a contralateral breast cancer on study imaging following randomization will remain in the study),
* Known pregnancy or lactating female,
* Inability to complete the study or required follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients upstaged to Stage IV disease | Within 30 days from date of randomization
  Proportion of patients upstaged to Stage IV disease as a result of the imaging study, between the groups

SECONDARY OUTCOMES:
Proportion of patients who receive multimodal therapy of curative intent | Within 12 months from date of randomization
Number of additional tests, such as imaging and biopsy, resulting from findings of study imaging | Within 12 months from date of randomization
Prognostic ability of PET SUV of the primary lesion on the pathological response rate to neo-adjuvant chemotherapy | Within 12 months from date of randomization
Disease Free Survival | From date of randomization to date of event, assessed up to 5 years
  Objectively defined local or distance recurrence or death
Overall Survival | From date of randomization to date of event, assessed up to 5 years
  Defined by all-cause mortality
Incremental economic analysis comparing the costs and outcomes of the treatment arms | Within 5 years from date of randomization
  Utility values will be collected using the EQ-5D Health Utility Questionnaire and converted to quality adjusted life years (QALYs) by considering Overall Survival. Direct medical resources (i.e. tests, complications, hospitalizations, clinic visits, emergency dept., etc.) will be obtained. Costs ($CAN2016) for each resource identified and utilized will be determined. Finally, an incremental cost-utility analysis will be calculated comparing the 2 randomized arms to generate an incremental cost per QALY outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Dayes, MD, Principal Investigator — Juravinski Hospital and Cancer Centre; Andrea Eisen, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Ralph George, MD, Principal Investigator — St. Michael's Hospital, CIBC Breast Centre; Ur Metser, MD, Principal Investigator — Princess Margaret Hospital, Canada; Mark Levine, MD, Study Director — Ontario Clinical Oncology Group (OCOG)
Locations (6):
- Canada (6):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metser U, Ali Mirshahvalad S, Dayes IS, Parpia S, Levine MN. 18F-FDG PET/CT of Oligometastatic Disease in Locally Advanced Breast Cancer: PETABC Trial Post Hoc Analysis. Radiology. 2025 Aug;316(2):e243788. doi: 10.1148/radiol.243788. PMID 40762843
- [Derived] Dayes IS, Metser U, Hodgson N, Parpia S, Eisen AF, George R, Blanchette P, Cil TD, Arnaout A, Chan A, Levine MN. Impact of 18F-Labeled Fluorodeoxyglucose Positron Emission Tomography-Computed Tomography Versus Conventional Staging in Patients With Locally Advanced Breast Cancer. J Clin Oncol. 2023 Aug 10;41(23):3909-3916. doi: 10.1200/JCO.23.00249. Epub 2023 May 26. PMID 37235845